CLINICAL TRIAL: NCT05178537
Title: Cross-sectional Study of 1200 Recreational Athletes With Former or Current Use of Performance and Image Enhancing Drugs, Focusing on Androgenic Anabolic Steroid
Brief Title: Cross-sectional Study of 1200 Recreational Athletes With Former or Current Use of Androgenic Anabolic Steroids
Acronym: FIDODK/BIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jan Frystyk (Other)
Responsible Party: Sponsor-Investigator, Jan Frystyk, Clinical professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: BICAAS01
Record Dates: First submitted 2021-12-13; First posted 2022-01-05 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Morbidity; Androgen Deficiency; Heart Failure
Keywords: cardiovascular morbidity; doping; anabolic steroids
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AAS users: current og previous use of AAS
  Interventions: Other: AAS users

INTERVENTIONS:
Other: AAS users — no intervention
  Other Names: no intervention

SUMMARY:
Overarching aim of project Performance and image enhancing drugs (PIEDs) are pharmacological agents acquired illicitly to improve physical strength and endurance as well as to obtain a leaner and more muscular appearance. Androgenic anabolic steroids (AAS) are the most frequently used PIED and include testosterone and its synthetic derivatives. However, PIEDs also include other hormones, e.g. growth hormone (GH), insulin-like growth factor I (IGF-I), glucocorticoids, insulin and thyroxin.

Originally, the use of PIEDs was predominately restricted to elite athletes. However, today most users of PIEDs are recreational athletes. In USA, the prevalence of recreational PIED users (three million) exceeds the prevalence of type 1 diabetes. This appears to be the same in Denmark, where the estimated prevalence of recreational users of PIEDs is 44,000, compared to approximately 30,000 patients with type 1 diabetes. The access to AAS is easy due to the unregulated and illicit sale on the internet. Furthermore, PIED use is common in the young population with possible detrimental effects on future health and well-being.

PIEDs are linked to premature death and a wide spectrum of somatic and psychological disorders. However, clinical data on the use of PIEDs is currently limited. Randomized trials of PIEDs are unethical as this would require administration of potentially harmful supra-physiological doses of hormones and this is the rationale behind our proposal to perform an observational study.

With this project the investigators propose to

a) Perform a cross-sectional nationwide study of current and former users of PIEDs (N=1200), focusing on AAS. In particular, the investigators will pay attention to:

1. Preclinical cardiovascular disease
2. Psychological well-being, aggression and quality of life
3. Biomarkers of ageing
4. Body composition and muscle strength b) Establish a nationwide biobank containing blood, urine and hair samples from current and former users of PIEDs.

DETAILED DESCRIPTION:
Performance and image enhancing drugs (PIEDs) are pharmacological agents acquired illicitly to improve physical strength and endurance as well as to obtain a leaner and more muscular appearance. Androgenic anabolic steroids (AAS) are the most frequently used PIED and include testosterone and its synthetic derivatives. However, PIEDs also include other hormones, e.g. growth hormone (GH), insulin-like growth factor I (IGF-I), glucocorticoids, insulin and thyroxin.

Originally, the use of PIEDs was predominately restricted to elite athletes. However, today most users of PIEDs are recreational athletes. In USA, the prevalence of recreational PIED users (three million) exceeds the prevalence of type 1 diabetes. This appears to be the same in Denmark, where the estimated prevalence of recreational users of PIEDs is 44,000, compared to approximately 30,000 patients with type 1 diabetes. The access to AAS is easy due to the unregulated and illicit sale on the internet. Furthermore, PIED use is common in the young population with possible detrimental effects on future health and well-being.

PIEDs are linked to premature death and a wide spectrum of somatic and psychological disorders. However, clinical data on the use of PIEDs is currently limited. Randomized trials of PIEDs are unethical as this would require administration of potentially harmful supra-physiological doses of hormones and this is the rationale behind our proposal to perform an observational study.

With this project the investigators propose to

a) Perform a cross-sectional nationwide study of current and former users of PIEDs (N=1200), focusing on AAS. In particular, the investigators will pay attention to:

1. Preclinical cardiovascular disease
2. Psychological well-being, aggression and quality of life
3. Biomarkers of ageing
4. Body composition and muscle strength b) Establish a nationwide biobank containing blood, urine and hair samples from current and former users of PIEDs.

   Study population Inclusion criteria

   • Recreational athletes (≥18 years of age) with current or former use of PIEDs, including AAS for ≥ 3 months

   Exclusion criteria

   • Severe psychiatric or somatic diseases which makes it impossible to give informed consent or comply with the investigatory program

   Estimated number of participants over 3 years are N=1200. Participants are recruited using social media groups, newspapers, posters in fitness centers and at general practitioners. Recruitment is performed in collaboration with Anti Doping Denmark.

   Investigations Patient reported outcomes (PRO) Bio impedance Muscle strength measurement Clinical examination Medical history and socioeconomic status Blood and urine samples Ultrasound of the carotid artery and aorta Echocardiography and ECG

   CHANGE IN PRIMARY ENDPOINT

   Amendment - modification of the description of the primary end-point: January 16, 2024.

   This clinical study is descriptive: It aims to describe the cardiovascular and mental health status of recreational athletes using anabolic androgenic steroids. As such, no strict statistical power calculations were performed.

   Originally, the primary endpoint was ultrasound-detected calcifications of aorta using a 3.5 mHz transducer.

   However, due to body size of the anabolic androgenic steroid using participants, the results have appeared not to be reliable. This became evident after the pilot study, which has included 120 recreational athletes.

   Consequently, the primary endpoint was modified to ultrasound-determined plaques of the carotid and the femoral arteries; i.e. North and South of the abdominal aorta.

ELIGIBILITY:
Inclusion Criteria:

* Recreational athletes (≥18 years of age) with current or former use of PIEDs, including AAS for ≥ 3 months

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recreational athletes (≥18 years of age) with current or former use of PIEDs, including AAS for ≥ 3 months
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound aorta | 1 day (Only one timepoint as the study is cross sectional)
  calcifications
Ultrasound of the carotid arteries and the femoral arteries | 1 day (Only one timepoint as the study is cross sectional)
  calcifications

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frystyk, Principal Investigator — Odense University Hospital
Locations (1):
- Jan Frystyk, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buhl LF, Lehmann Christensen L, Diederichsen A, Lindholt JS, Kistorp CM, Glintborg D, Andersen M, Frystyk J. Impact of androgenic anabolic steroid use on cardiovascular and mental health in Danish recreational athletes: protocol for a nationwide cross-sectional cohort study as a part of the Fitness Doping in Denmark (FIDO-DK) study. BMJ Open. 2024 May 7;14(5):e078558. doi: 10.1136/bmjopen-2023-078558. PMID 38719280